CLINICAL TRIAL: NCT02946489
Title: Facilitating the Behavioral Treatment of Cannabis Use Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Elias Dakwar, research psychiatrist, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 7355; K24DA029647 (NIH)
Record Dates: First submitted 2016-10-20; First posted 2016-10-27 (Estimated); Results first posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-01

CONDITIONS: Cannabis Dependence
Keywords: cannabis; mindfulness based relapse prevention; motivational enhancement therapy
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant
Masking Description: Open label single-blind trial, with participants given the impression they may get any of several medications.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CI-581a+MET+MBRP (Experimental): Administration of CI-581a during wk 2 and possibly at wk 3 or 4 at 0.71 mg/kg in the context of a 2 wk course of MET followed by a 4 wk course of MBRP
  Interventions: Drug: CI-581a

INTERVENTIONS:
Drug: CI-581a — CI-581a will be administered in wk2 and potentially in wk 3 or 4.

SUMMARY:
Cannabis use disorders remain a significant public health problem. The pharmacological facilitation of behavioral treatment represents a promising strategy for addressing disordered cannabis use. Cannabis use disorders are recognized to be associated with various vulnerabilities that complicate the course of treatment and that may be amenable to glutamate modulators. The purpose of this single blind open-label trial is to test the feasibility of administering glutamate modulators in conjunction with motivational enhancement therapy (MET) and mindfulness based relapse prevention (MBRP) for cannabis use disorders.

DETAILED DESCRIPTION:
Individuals diagnosed with cannabis dependence will receive one or two infusions of glutamate modulators during week 2 and week 3 or 4. The participants will also receive 2-week course of MET and 4-week course of MBRP. Participants will meet with staff twice weekly, except for week 2 and potentially week 3 or 4 during which participants will present to the clinic three times. Clinic visits include MET sessions, MBRP sessions, psychiatric monitoring, assessments, and study procedures (e.g., medication administration).

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for cannabis dependence, with at least 5 days of use per week over the past 30 days and displaying at least one positive utox during screening
* Physically healthy
* No adverse reactions to study medications
* 21-60 years of age
* Capacity to consent and comply with study procedures
* Seeking treatment

Exclusion Criteria:

* Meets DSM IV criteria for current major depression, bipolar disorder, schizophrenia, any psychotic illness, including substance-induced psychosis, and current substance-induced mood disorder.
* Physiological dependence on another substance requiring medical management, such as alcohol, opioids, or benzodiazepines, excluding caffeine, and nicotine.
* Pregnant, interested in becoming pregnant, or lactating
* Delirium, Dementia, Amnesia, Cognitive Disorders, or dissociative disorders
* Current suicide risk or a history of suicide attempt within the past 2 years
* On psychotropic or other medication whose effect could be disrupted by participation in the study
* Recent history of significant violence (past 2 years).
* Heart disease as indicated by history, abnormal ECG, previous cardiac surgery.
* Unstable physical disorders which might make participation hazardous such as end-stage AIDS, hypertension (>140/90), anemia, pulmonary disease, active hepatitis or other liver disease (transaminase levels < 2-3 X the upper limit of normal will be considered acceptable), or untreated diabetes
* Previous history of misuse of study medications
* BMI > 35, or a history of undocumented obstructive sleep apnea
* First degree relative with a psychotic disorder (bipolar disorder with psychotic features, schizophrenia, schizoaffective disorder, or psychosis NOS)

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elias Dakwar, MD, Principal Investigator — Columbia University
Locations (1):
- NYSPI, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CI-581a+MET+MBRP
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CI-581a+MET+MBRP
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 4
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Cannabis Abstinence or Significant Reduction in Cannabis Use
Description: Percentage of participants with cannabis abstinence or significant reduction in cannabis use by end of study. Significant reduction in cannabis use was defined as: At least 50% reduction in cannabis use between pre-infusion and end of 6 week study.
Time Frame: At Week 6 (End of study)
Measure: Count of Participants; unit: Participants
Arm/Group | CI-581a+MET+MBRP
Number analyzed (Participants) | 8
Participants | 7

2. Secondary Outcome: Confidence in Abstaining From Cannabis
Description: Change in confidence in abstaining from cannabis as measured by the DCQ (Drug-Taking Confidence Questionnaire). DCQ is a scale from 0 to 100, with higher values indicating greater confidence in one's ability to abstain from cannabis.
Time Frame: Change between pre-infusion and end of 6 week study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CI-581a+MET+MBRP
Number analyzed (Participants) | 8
units on a scale | 42.8125 (27.56283)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the study period (6 weeks)
Arm/Group | CI-581a+MET+MBRP
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT02946489/Prot_000.pdf